CLINICAL TRIAL: NCT05868226
Title: PRE-Investigation of Serial Studies to Predict Your Therapeutic Response With Imaging And moLecular Analysis: A Phase I/Ib Platform Trial
Brief Title: PRE-I-SPY Phase I/Ib Oncology Platform Program
Acronym: PRE-I-SPY-PI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: QuantumLeap Healthcare Collaborative (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-SPY-P1
Record Dates: First submitted 2022-04-22; First posted 2023-05-22 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: HER2-positive Breast Cancer; Metastatic Cancer; Metastatic Breast Cancer; Metastatic; HER2-positive Metastatic Breast Cancer; HER2 Mutation-Related Tumors; HER-2 Protein Overexpression; HER2-negative Breast Cancer; Triple Negative Breast Cancer; HR Positive; Hormone Receptor-positive Breast Cancer; Estrogen Receptor Positive Tumor; Progesterone Receptor-positive Breast Cancer; Hormone Receptor Negative Breast Carcinoma; Solid Tumor; Solid Tumor, Adult; Solid Carcinoma; HER2 Low Breast Cancer; HER2 Low Breast Carcinoma; ER Positive Breast Cancer; PR-positive Breast Cancer
Keywords: I-SPY Trials; Quantum Leap Healthcare Collaborative; QLHC; I-SPY; I-SPY2; I-SPY1; PRE-ISPY; PRE-I-SPY; I-SPY Phase 1; I-SPY Phase 1b; I-SPY-P1; ISPY; ISPYP1; I-SPY Phase 1 Platform; ISPY2; ISPY1; Phase 1 Platform; Phase 1 Oncology Platform; T-DXd naive; PRE1; PRE2; PRE3; PRE; PRE-I-SPY Phase 1; PRE-I-SPY Phase 1b; ALX148; T-DXd; Enhertu; Zanidatamab; Tucatinib; Ziihera; Tukysa; Evorpacept; QL
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — ALX148; zanidatamab; tucatinib

STUDY DESIGN:
Intervention Model Description: This is an open-label, multi-site, multi-arm platform study, where each drug regimen arm may have different study designs and eligibility. In particular, dose finding parts may employ different designs (e.g., 3+3, Bayesian Optimal Interval Design [BOIN], continual reassessment method [CRM], etc.) for each arm in the PRE-I-SPY program. See each arm for specific study model details.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRE1 ALX148 (Evorpacept) + Fam-Trastuzumab Deruxtecan-Nxki (T-DXd, Enhertu®) (Experimental): The combination of T-DXd and ALX148 aims to explore the anti-tumoral effects of trastuzumab, of the topoisomerase inhibitor DXd and of the CD47-blocking agent ALX148. The rationale for this combination is that ALX148 is hypothesized, based on preclinical data, to facilitate antibody-dependent cellular phagocytosis (ADCP) of HER2 expressing (>HER2 1+) breast cancer binding T-DXd while cancer cell intrinsic or bystander cytotoxicity of T-DXd will result in the release of neoantigens promoting immune mediated antitumor activity in the tumor microenvironment.
  Interventions: Drug: ALX148; Drug: Fam-Trastuzumab Deruxtecan-Nxki
- PRE2 Zanidatamab (Ziihera®, ZW25, zani) + Tucatinib (TUKYSA®) (Experimental): Zanidatamab is a bispecific IgG1-like antibody directed against two distinct HER2 epitopes. It induces formation of receptor clusters and internalization resulting in downregulation. It also inhibits growth factor-dependent and -independent tumor cell proliferation and potently activates ADCC, ADCP, and CDC. FDA approved for metastatic HER2+ bile duct cancer.
  Tucatinib is a highly selective, small molecule tyrosine kinase inhibitor (TKI) of HER2 compared to other TKI's (i.e., EGFR). It is well tolerated, crosses the blood brain barrier and can treat CNS disease. FDA approved for HER2+ breast cancer.
  Given the promising clinical data for each of these drugs which have different mechanisms, the effect of zanidatamab after T-DXd (Enhertu®) in breast cancer patients, and the favorable toxicity profile of both drugs, we hypothesize that the combination of tucatinib and zanidatamab will be well tolerated and more efficacious than either drug alone for the treatment of HER2+ breast cancer.
  Interventions: Drug: Zanidatamab; Drug: Tucatinib

INTERVENTIONS:
Drug: ALX148 — CD47 Inhibitor: A fusion protein containing a high affinity engineered D1 domain of human signal regulatory protein alpha (SIRPα) variant 1 (v1) genetically linked to a modified and inactive Fc domain of human immunoglobulin (Ig) G1.
  Other Names: Evorpacept
  Arms: PRE1 ALX148 (Evorpacept) + Fam-Trastuzumab Deruxtecan-Nxki (T-DXd, Enhertu®)
Drug: Fam-Trastuzumab Deruxtecan-Nxki — Antibody-drug conjugate (ADC): A recombinant humanized anti-human HER2 IgG1 monoclonal antibody, conjugated with linker to a Topoisomerase I inhibitor
  Other Names: Enhertu; T-DXd
  Arms: PRE1 ALX148 (Evorpacept) + Fam-Trastuzumab Deruxtecan-Nxki (T-DXd, Enhertu®)
Drug: Zanidatamab — Bispecific HER2 antibody: A humanized, bispecific, immunoglobulin G isotype 1 (IgG1)-like antibody directed against the juxtamembrane extracellular domain (ECD4) and the dimerization domain (ECD2) of human epidermal growth factor receptor 2 (HER2).
  Other Names: ZW25; zani; Ziihera
  Arms: PRE2 Zanidatamab (Ziihera®, ZW25, zani) + Tucatinib (TUKYSA®)
Drug: Tucatinib — Small molecule tyrosine kinase inhibitor (TKI) of HER2 (oral drug).
  Other Names: TUKYSA
  Arms: PRE2 Zanidatamab (Ziihera®, ZW25, zani) + Tucatinib (TUKYSA®)

SUMMARY:
I-SPY Phase I/Ib (I-SPY-P1) is an open-label, multisite platform study designed to evaluate single agents or combinations in a metastatic treatment setting that may be relevant for breast cancer patients with the overall goal of moving promising drug regimens into the I-SPY 2 SMART Design Trial (NCT01042379) and/or other oncology-based trials in a timely manner.

DETAILED DESCRIPTION:
The PRE-I-SPY/I-SPY-P1 study is a platform trial with multiple ongoing drug regimen arms. In most cases, the treatment arm will have a dose-finding group (Part 1) and a dose-expansion group (Part 2). Eligibility criteria will vary according to the experimental regimen. Participant eligibility may vary according to the arm or the part within the study arm, including with respect to diagnosis. Arms could include participants diagnosed with certain solid tumors or specifically with breast cancer. Arms may restrict enrollment to a certain molecular pathway abnormality or histologic diagnosis. The trial allows for various study arm designs, with the goal to complete analysis of a study arm in 12 to 18 months.

ELIGIBILITY:
General Inclusion Criteria (GIC):

* GIC1: The participant must have ability to understand and willingness to provide signed written informed consent prior to any study related assessments and procedures and for collection of archival FFPE blocks (freshly cut 14 unstained tumor slides would be acceptable).
* GIC2: Age ≥ 18 years at the time of signing the informed consent
* GIC3: Gender: Male or female (premenopausal and postmenopausal)
* GIC4: ECOG performance status Grade 0-2
* GIC5: Estimated life expectancy > 12 weeks at the start of investigational medicinal product (IMP) treatment.
* GIC6: Adequate organ function, evidenced by the following laboratory results within 30 days of the start of IMP:

  * Absolute neutrophil count ≥ 1,500/mm3
  * Platelet count ≥ 100,000/mm3
  * Hemoglobin ≥ 9.0 g/dL with no blood transfusion in the past 28 days
  * Total bilirubin ≤ 1.5 x the upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x ULN
  * Estimated Creatinine clearance (using Cockcroft-Gault formula) ≥ 60 mL/min for small molecules and >30 mL/min for monoclonal antibodies unless otherwise specified in the Arm Specific Eligibility.

These cut-off values may be modified with supporting data for specific drug regimens.

* GIC7: Non-Pregnant: Serum or urine pregnancy test must be negative within 14 days of IMP treatment start in women of childbearing potential. Pregnancy testing does not need to be pursued in patients who are judged as postmenopausal before enrollment, or who have undergone bilateral oophorectomy, total hysterectomy, or bilateral tubal ligation. If male, they must agree to refrain from donating sperm during treatment.
* GIC8: Contraception: Women of childbearing potential and men must be willing to use adequate contraception for the duration of protocol treatment. Additional information regarding contraception for the specific treatment arm will be added to the drug arm description. Adequate contraception is defined as one highly effective form (i.e., abstinence, (fe)male sterilization) OR two effective forms (e.g., non-hormonal IUD and condom / occlusive cap with spermicidal foam / gel / film / cream / suppository).
* GIC9: Prior therapy effects: Resolution of all acute toxic effects of prior therapy, including radiotherapy, to grade ≤1 and neuropathy to grade ≤2 (except toxicities not considered a safety risk for the patient) and recovery from surgical procedures.
* GIC10: Participant compliance: Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Additional arm specific inclusion criteria as needed by drug arm regimen

General Exclusion Criteria (GEC):

* GEC1: Wash out periods: No other anticancer therapy within the following periods:

  * chemotherapy or investigational agents, 3 weeks
  * mitomycin C and nitrosoureas, 6 weeks
  * radiotherapy, 3 weeks
  * targeted therapy, 2 weeks
  * MAbs, ADCs, and immunotherapy, 3 weeks
  * endocrine therapy, no washout needed
* GEC2: Concurrent therapy with other Investigational Products.
* GEC3: Prior history of drug/regimen hypersensitivity: History of infusion-related reactions and/or hypersensitivity to IMP or excipients of the study drug/drugs which led to permanent discontinuation of the treatment.
* GEC4: Uncontrolled intercurrent illness including (active infection, diabetes, pulmonary embolism in the past 6 months, or psychiatric illness/social situations that would limit compliance with study requirements).
* GEC5: Cardiovascular disease: History (within 6 months prior to start IMP) of clinically significant cardiovascular disease such as unstable angina, congestive heart failure (CHF), myocardial infarction, uncontrolled hypertension, cardiac arrhythmia requiring medication, or baseline corrected QT by Fridericia's formula (QTcF) length > 470 msec for men and women. The QTcF cut-off value may be modified with supporting data for specific drug regimens.
* GEC6: CNS tumoral spread: Active uncontrolled/symptomatic central nervous system cancer/spinal cord compression. Previously treated and clinically stable lesions, as per Investigator's judgment, are permitted. Newly discovered asymptomatic lesions that are not life threatening and do not require urgent local treatment to ensure patient safety, after consultation with study regimen chaperones, may be permitted.
* GEC7: Liver disease: Patients with clinically significant history of liver disease, including viral or other known hepatitis, current alcohol abuse, or cirrhosis.
* GEC8: Recent major surgery within 4 weeks prior to start IMP treatment
* GEC9: Pregnancy or breastfeeding
* GEC10: Individuals accommodated in an institution because of regulatory or legal order; prisoners or participants who are legally institutionalized.
* GEC11: Other conditions, which in the opinion of the investigator, would compromise the safety of the patient or the patient's ability to complete the study.
* GEC12: Concomitant malignancies: A diagnosis of a malignancy in the 2 years prior to starting study treatment other than the disease under study. Exceptions include indolent or definitively treated malignancy not expected to require treatment during the study, affect the safety of subjects, or affect the endpoints of the trial.
* Additional arm specific exclusion criteria as needed by drug arm regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events related to the treatment | Start of treatment to 30 days post treatment (estimated 12 -18 months)
  Evaluate the number of adverse events related to the treatment according to the current version of CTCAE during the trial.
Incidence of Dose Limiting Toxicities (DLTs) at each dose level | DLT observation period: Start of treatment to 21 days (Cycle 1)
  To determine the safety and tolerability of new agents/regimens in participants with certain advanced solid tumors and breast cancer. DLT rate (number of participants who experience a protocol defined DLT/total number of DLT cohort participants at that dose).
Maximum Tolerated Dose (MTD) | Start of treatment to the date of last participant at end of DLT observation period at highest dose level (estimated 6 months)
  The maximum dose level (mg/kg) which is not eliminated.
Recommended Phase 2 Dose (RP2D) | Start of treatment to the date of last participant at highest dose level (estimated 6 months)
  Using all available data, computation of RP2D (mg/kg), which may not be the MTD.
Overall Response Rate (ORR) | Start of treatment to 12 months
  To obtain preliminary efficacy data of the new agents/regimens in participants with certain advanced solid tumors and breast cancer.
Duration of Response (DOR) | Start of treatment to 12 months
  To obtain preliminary efficacy data of the new agents/regimens in participants with certain advanced solid tumors and breast cancer.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) - descriptive | Start of treatment to 12 months
  To provide descriptive assessment of Progression Free Survival (PFS) of the new agents/regimens with certain advanced solid tumors and breast cancer
Clinical Benefit Rate (CBR) at 6 months | Start of treatment to 6 months
  To obtain preliminary Clinical Benefit Rate (CBR) at 6 months of participants treated with the new agents/regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Paula R Pohlmann, MD, MSc, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (7):
- United States (7):
  - The University of Alabama at Birmingham O'Neal Comprehensive Cancer Center, Birmingham, Alabama
  - Moffitt Cancer Center, Tampa, Florida
  - The University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois
  - UChicago Medicine Comprehensive Cancer Center at Silver Cross Hospital, New Lenox, Illinois
  - UChicago Medicine Orland Park, Orland Park, Illinois
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - The University of Texas MD Anderson Cancer Center, Houston, Texas